CLINICAL TRIAL: NCT01695460
Title: A Randomized, Parallel, Double-blind, Placebo-controlled Study of Vitamin D as Prophylactic Treatment for Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: CCBR Aalborg A/S, Aalborg, Denmark (Unknown); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Parisa Gazerani, Associate Professor, Pharm D, PhD, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-20120052; Projekt #831302 (Other Grant/Funding Number: Det Frie Forskningsråd)
Record Dates: First submitted 2012-09-25; First posted 2012-09-28 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Migraine According to International Headache Society (IHS) Criteria (ICHD-II)
Keywords: Migraine; Vitamin D
MeSH Terms: conditions — Migraine Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): The active treatment consists of vitamin D and is given in tablets of the brand D3 Vitamin ®, supplied by D3 Pharmacy Ltd., Bispensgade 22, 9000 Aalborg.
  The tablets contain the vitamin D in the form of vitamin D3, also known as cholecalciferol.
  D3 Vitamin ® consists of small white tablets, which are easy to swallow.
  D3 Vitamin ® contains 25 micrograms vitamin D3 (colecalciferol) per tablet, equivalent to 1000 IU (International Units).
  Tablet Excipients: Cellulose, dicalcium phosphate, magnesium stearate, silicon dioxide and talc. Vitamin D3 ® contains no gluten, soy, gelatin or other animal products.
  Interventions: Drug: D3 Vitamin ®
- Placebo (Placebo Comparator): Placebo tablets to match D3 Vitamin ®, were produced. They are identical to the D3 Vitamin ® in appearance, ie small white tablets. These tablets do not have a therapeutic effect. Placebo tablets produced and delivered by D3 Pharmacy Ltd., Bispensgade 22, 9000 Aalborg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D3 Vitamin ® — Vitamin D and placebo supplied as tablets in containers of 124. The containers must be kept in dry and not too hot environment.
  All subjects randomized to vitamin D, will receive 100 micrograms of vitamin D3/day, equivalent to 4000 IU. Vitamin D is administered orally 1 time a day with breakfast.
  Other Names: D3 Vitamin ®, supplied by D3 Pharmacy Ltd
  Arms: Vitamin D
Drug: Placebo
  Other Names: Placebo tablets to match D3 Vitamin ®, produced by D3 Pharmacy Ltd
  Arms: Placebo

SUMMARY:
The trial is primarily designed to investigate whether treatment with vitamin D may influence migraine in a placebo-controlled, blinded study. The hypothesis is that vitamin D may serve as a prophylactic treatment of migraine. The hypothesis is tested by examining the changes in the pain and symptom patterns associated with migraine by treatment with Vitamin D, by means of quantitative sensory testing, diaries and blood samples for measurement of vitamin D. Other pain biomarkers are also measured to evaluate whether the levels of these biomarkers in the blood is changed by the treatment with vitamin D. The hypothesis here is that levels of those biomarkers will change following the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65, migraine must have occurred before the age of 50 years.
* Diagnosed migraine according to International Headache Society (IHS) criteria (ICHD-II)

Exclusion Criteria:

* Other neurological or neurodegenerative disorders
* Medical conditions that may interfere with the result - violent head trauma, stroke, transient ischemic attacks
* Musculoskeletal or mental illness
* Addictive or previous addictive behavior defined as the abuse of cannabis, opioids or other drugs
* Inability to cooperate
* Pregnancy or breastfeeding, including women trying to conceive
* Use of vitamin D supplementation> 10μg
* In treatment with digoxin or thiazide
* Patients with osteoarthritis, as they are taking or have taken vitamin D supplements
* Patients with pre-existing hypercalcemia as vitamin D supplements are contraindicated in these patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The number of migraine attacks | every 4 weeks
  The primary endpoint is the frequency of migraine attacks. This is estimated from the subjects' listing of attacks in the form of diaries. This is assessed as the number of migraine attacks per 4 weeks (28 days).

SECONDARY OUTCOMES:
Evaluation of pain during migraine attacks | every 4 weeks
  Evaluation of pain during migraine attacks carried out by the subjects themselves by completing diaries. The diaries trial participants evaluate the pain intensity during an attack using a 1-3 scale, where 1 is mild pain, 2 is moderate pain, and 3 severe pain.
Hypersensitivity | Baseline and every 4 weeks
  allodynia and hyperalgesia (hypersensitivity) assessed by standardized questions about the sensitivity of the skin associated with migraine.
Migraine Symptoms | every 4 weeks
  Migraine Symptoms, including aura, nausea, light and sound sensitivity are also assessed by trial participants using diaries.
Quantitative Sensory Testing | Every 4 weeks
  Pain Pressure Threshold and temporal summation are measured.
Measuring levels of a biomarker. Changes in the levels of these biomarkers. | Baseline and after 6 months treatment (end of trial)
  Changes in the levels of these biomarkers are measured:
  25(OH)D, 1,25(OH)D, GFAP, S100B, CGRP,Glutamate, Serotonin, Prostaglandin E2

OTHER OUTCOMES:
Quality of life | Every 28 days
  HIT-6 (Headache Impact Test)

CONTACTS AND LOCATIONS:
Overall Officials: Parisa Gazerani, Pharm D, PhD, Study Chair — Aalborg University
Locations (2):
- Denmark (2):
  - CCBR Aalborg A/S, Aalborg
  - Aalborg University, Aalborg

REFERENCES:
- [Derived] Gazerani P, Fuglsang R, Pedersen JG, Sorensen J, Kjeldsen JL, Yassin H, Nedergaard BS. A randomized, double-blinded, placebo-controlled, parallel trial of vitamin D3 supplementation in adult patients with migraine. Curr Med Res Opin. 2019 Apr;35(4):715-723. doi: 10.1080/03007995.2018.1519503. Epub 2018 Sep 28. PMID 30182753